CLINICAL TRIAL: NCT00545831
Title: Prevention of Central Veinous Device Related Sepsis Relapse With Taurolidine in Patients on Parenteral Nutrition in Long-term Home
Brief Title: Effect of Taurolidin on Prevention of Bloodstream Infection
Acronym: Nutrilock
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of recruitment
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2006/100/HP; 2007-A00618-45
Record Dates: First submitted 2007-10-16; First posted 2007-10-17 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Sepsis
Keywords: Home Parenteral Nutrition; Sepsis Prevention; Central Venous Catheters; Taurolidine
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Use of taurolidine in prevention of bloodstream infection related to central venous access
  Interventions: Device: Taurolidine
- B (Placebo Comparator): Use of Physiologic Serum to compare to arm A
  Interventions: Device: Physiologic Serum

INTERVENTIONS:
Device: Taurolidine — 2 mL of taurolidine instillate on the intravascular catheter after each parenteral nutrition session for a duration of 6 months
  Arms: A
Device: Physiologic Serum — 2 mL of physiologic serum instillate on the intravascular catheter after each parenteral nutrition session for a duration of 6 months
  Arms: B

SUMMARY:
Home parenteral nutrition (HPN) is a validated technique for patients with various intestinal disease leading to chronic malabsorption or obstruction, whatever the aetiology. Intravascular catheter-related bloodstream infections (CRBSI) is the more frequent complication of patients with HPN and an important cause of morbidity and mortality in these patients. Moreover, CRBSI often recur after a first treatment of the catheter with a combination of an antibiotic lock on the catheter and systemic intravenous antibiotics. In more than 50 % of the cases, another CRBSI will occur in a median delay of 5 months.

The aim of the study is to evaluate the efficacy of a taurolidine lock secondary prophylaxis on CRBSI recurrence in HPN patients.

Study population is separated in 2 groups, the first one receiving the Taurolock and the second one receiving a placebo. This is a randomized double-blind six-month study.

ELIGIBILITY:
Inclusion Criteria:

* Age superior to 18 years
* Home parenteral nutrition on tunnelized central venous catheters
* Bloodstream infection confirmed by differential hemocultures
* Informed consent form signed
* Negative B-HCG test

Exclusion Criteria:

* Subject unable to give his informed consent
* Pregnancy
* Subject who have a two or three-way catheter, or a non-tunnelized central venous catheter
* Hospital related infection
* Central venous catheters placed since less than 15 days
* Neutropenia < 500 PNN/mm3
* Fungal Infection, polymicrobial who need ablation of the central venous catheters
* No-response to clinical treatment of the Infection
* Septic thrombophlebitis
* Chemotherapy ongoing
* On going malignancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2007-10; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Number of recurrence of catheter-related infection in each group | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Lecleire, MD, Principal Investigator — University Hospital, Rouen
Locations (7):
- France (7):
  - APHP Beaujon Hospital, Clichy
  - UH of Grenoble, Grenoble
  - UH of Lille, Lille
  - UH of Lyon, Lyon
  - UH of Nice, Nice
  - University Hospital of Rouen, Rouen
  - UH of Toulouse, Toulouse